CLINICAL TRIAL: NCT00502944
Title: Optimizing Strategies for Universal HIV Testing (The USHER Trial)
Brief Title: Two Approaches to Routine HIV Testing in a Hospital Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rochelle Walensky, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R01MH073445 (NIH); R01MH073445 (NIH); DAHBR 9A-ASPQ
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: HIV Infections
Keywords: HIV; Testing; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counselor-based HIV screening (Experimental)
  Interventions: Behavioral: Counselor-based HIV screening
- Emergency staff member-based HIV screening (Active Comparator)
  Interventions: Behavioral: Emergency staff member-based HIV screening

INTERVENTIONS:
Behavioral: Counselor-based HIV screening — Participants will undergo oral HIV screening by HIV counselor and, if positive, further study visits for up to 6 months
  Arms: Counselor-based HIV screening
Behavioral: Emergency staff member-based HIV screening — Participants will undergo oral HIV screening by emergency staff member and, if positive, further study visits for up to 6 months
  Arms: Emergency staff member-based HIV screening

SUMMARY:
This study will compare the effectiveness of two different approaches to providing routine HIV counseling, testing, and referral services in an urban hospital emergency department setting.

DETAILED DESCRIPTION:
About 25% of HIV infected people do not know that they are infected. These people lack medical care that could prolong their lives and access to counseling services that could prevent further spread of HIV. With so many people unaware of their HIV status, there is a clear need for more readily available HIV counseling, testing, and referral services throughout the United States. The Centers for Disease Control and Prevention (CDC) recommends routine HIV testing in U.S. hospitals in which HIV infected patients make up at least 1% of the total patient population for that hospital. However, routine HIV testing in such hospitals is rarely carried out, which might be because the CDC has not specified who should perform routine HIV testing. The purpose of this study is to compare the effectiveness of two different approaches to providing routine HIV counseling, testing, and referral services in an urban hospital emergency department setting. One approach will be led by an HIV counselor, and the other approach will be led by an emergency department staff member. For both approaches, the study will evaluate to what extent patients accept HIV testing, how well follow-up care is established, and the cost-effectiveness of the approach.

Participants in this study will include adults who visit Brigham and Women's Hospital emergency department in Boston, Massachusetts. Participants will be randomly assigned to a counselor versus provider and will be asked to fill out a questionnaire while waiting in the emergency room. The questionnaire will be anonymous. Participants will then be offered an oral rapid HIV test. Test results will be available in about 20 minutes and will be provided to participants by either their assigned HIV counselor. Participants who test positive for HIV will be offered a more definitive blood test to confirm HIV infection. The blood test results will be available 2 weeks from testing, and participants must return to the hospital to get their test results. Participants who test positive for HIV will be offered counseling support and referral services by either their assigned HIV counselor or emergency department staff member. Follow-up care appointments will also be initiated at this time. For participants who test positive for HIV, the study will last about 6 months. There will be no follow-up visits for participants who do not test positive for HIV during their emergency room visit.

ELIGIBILITY:
Inclusion Criteria:

* Waiting to receive care in the Brigham and Women's Hospital emergency room
* English- or Spanish-speaking
* Enters the emergency room when an HIV counselor is available

Exclusion Criteria:

* An estimated severity index score of 1 or 2 who have mechanical ventilation or are not deemed alert, awake, and oriented to person, place and time by the triage nurse
* HIV infected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4855 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle P. Walensky, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Millen JC, Arbelaez C, Walensky RP. Implications and impact of the new US Centers for Disease Control and prevention HIV testing guidelines. Curr Infect Dis Rep. 2008 May;10(2):157-63. doi: 10.1007/s11908-008-0027-6. PMID 18462591
- [Background] Walensky RP, Freedberg KA, Weinstein MC, Paltiel AD. Cost-effectiveness of HIV testing and treatment in the United States. Clin Infect Dis. 2007 Dec 15;45 Suppl 4(Suppl 4):S248-54. doi: 10.1086/522546. PMID 18190295
- [Background] Ganguli I, Bassett IV, Dong KL, Walensky RP. Home testing for HIV infection in resource-limited settings. Curr HIV/AIDS Rep. 2009 Nov;6(4):217-23. doi: 10.1007/s11904-009-0029-5. PMID 19849965
- [Background] Reichmann WM, Losina E, Seage GR, Arbelaez C, Safren SA, Katz JN, Hetland A, Walensky RP. Does modality of survey administration impact data quality: audio computer assisted self interview (ACASI) versus self-administered pen and paper? PLoS One. 2010 Jan 15;5(1):e8728. doi: 10.1371/journal.pone.0008728. PMID 20090953
- [Background] Donnell-Fink L, Reichmann WM, Arbelaez C, Case AL, Katz JN, Losina E, Walensky RP. Patient satisfaction with rapid HIV testing in the emergency department. Ann Emerg Med. 2011 Jul;58(1 Suppl 1):S49-52. doi: 10.1016/j.annemergmed.2011.03.024. PMID 21684408
- [Background] Reichmann WM, Walensky RP, Case A, Novais A, Arbelaez C, Katz JN, Losina E. Estimation of the prevalence of undiagnosed and diagnosed HIV in an urban emergency department. PLoS One. 2011;6(11):e27701. doi: 10.1371/journal.pone.0027701. Epub 2011 Nov 16. PMID 22110730
- [Background] Pisculli ML, Reichmann WM, Losina E, Donnell-Fink LA, Arbelaez C, Katz JN, Walensky RP. Factors associated with refusal of rapid HIV testing in an emergency department. AIDS Behav. 2011 May;15(4):734-42. doi: 10.1007/s10461-010-9837-2. PMID 20978834
- [Result] Walensky RP, Arbelaez C, Reichmann WM, Walls RM, Katz JN, Block BL, Dooley M, Hetland A, Kimmel S, Solomon JD, Losina E. Revising expectations from rapid HIV tests in the emergency department. Ann Intern Med. 2008 Aug 5;149(3):153-60. doi: 10.7326/0003-4819-149-3-200808050-00003. PMID 18678842
- [Result] Arbelaez C, Block B, Losina E, Wright EA, Reichmann WM, Mikulinsky R, Solomon JD, Dooley MM, Walensky RP. Rapid HIV testing program implementation: lessons from the emergency department. Int J Emerg Med. 2009 Sep 1;2(3):187-94. doi: 10.1007/s12245-009-0123-x. PMID 20157472
- [Result] Arbelaez C, Wright EA, Losina E, Millen JC, Kimmel S, Dooley M, Reichmann WM, Mikulinsky R, Walensky RP. Emergency provider attitudes and barriers to universal HIV testing in the emergency department. J Emerg Med. 2012 Jan;42(1):7-14. doi: 10.1016/j.jemermed.2009.07.038. Epub 2009 Oct 14. PMID 19828278
- [Result] Walensky RP, Morris BL, Reichmann WM, Paltiel AD, Arbelaez C, Donnell-Fink L, Katz JN, Losina E. Resource utilization and cost-effectiveness of counselor- vs. provider-based rapid point-of-care HIV screening in the emergency department. PLoS One. 2011;6(10):e25575. doi: 10.1371/journal.pone.0025575. Epub 2011 Oct 12. PMID 22022415
- [Result] Walensky RP, Reichmann WM, Arbelaez C, Wright E, Katz JN, Seage GR 3rd, Safren SA, Hare AQ, Novais A, Losina E. Counselor- versus provider-based HIV screening in the emergency department: results from the universal screening for HIV infection in the emergency room (USHER) randomized controlled trial. Ann Emerg Med. 2011 Jul;58(1 Suppl 1):S126-32.e1-4. doi: 10.1016/j.annemergmed.2011.03.023. PMID 21684391
- [Derived] Ganguli I, Collins JE, Reichmann WM, Losina E, Katz JN, Arbelaez C, Donnell-Fink LA, Walensky RP. Missed opportunities: refusal to confirm reactive rapid HIV tests in the emergency department. PLoS One. 2013;8(1):e53408. doi: 10.1371/journal.pone.0053408. Epub 2013 Jan 8. PMID 23308216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from February 7, 2007 to July 9, 2008 at Brigham and Women's Hospital emergency department. Oral HIV testing was offered to eligible patients by either HIV counselors or emergency service assistants (existing members of emergency department personnel).
Groups:
- Counselor: Counselor-based HIV screening intervention where a dedicated HIV counselor does all the screening.
- Provider: Emergency staff member-based HIV screening intervention where an emergency staff member does all the screening.
Period: Overall Study
Arm/Group | Counselor | Provider
Started | 2446 | 2409
Completed | 1382 | 643
Not Completed | 1064 | 1766

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counselor | Provider | Total
Number analyzed (Participants) | 2446 | 2409 | 4855
Age Continuous [Mean (Standard Deviation); unit: years] | 37.1 (14) | 37.1 (14) | 37.1 (14)
Gender [Number; unit: participants] — Numbers within the gender category do not add up to total number randomized due to missing data/numbers.
  participants
    Female | 1585 | 1554 | 3139
    Male | 849 | 832 | 1681
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 938 | 928 | 1866
  Non-Hispanic Black | 526 | 546 | 1072
  Hispanic | 707 | 670 | 1377
  Asian/Asian-American | 66 | 59 | 125
  Native American/Alaskan Native | 12 | 8 | 20
  Multi-racial/Other | 176 | 164 | 340
  Missing | 21 | 34 | 55
Primary Language [Number; unit: participants]
  English | 1788 | 1807 | 3595
  Spanish | 483 | 448 | 931
  Other | 154 | 137 | 291
  Missing | 21 | 17 | 38
Education [Number; unit: participants]
  Less than High School | 310 | 310 | 620
  High School Degree | 566 | 575 | 1141
  Some College | 696 | 713 | 1409
  College Degree | 517 | 438 | 955
  Some Post-College/Graduate Degree | 342 | 347 | 689
  Missing | 15 | 26 | 41

OUTCOME MEASURES:

1. Secondary Outcome: Overall Rapid HIV Testing Rate
Description: We defined the overall rapid HIV testing rate as the number of participants tested for HIV using the rapid test among those randomized to potentially be tested in each arm.
Time Frame: Assess on day subject enrolled into the study
Population: Intention to treat analysis
Measure: Number; unit: participants
Arm/Group | Counselor | Provider
Number analyzed (Participants) | 2446 | 2409
participants | 1382 | 643
Statistical Analysis 1: Comparison: Counselor vs Provider; HIV test completed among patients randomized; Test type: Superiority or Other; p < 0.001, Chi-squared; Rate Difference (%) = 30, 95% CI 2-sided [27 to 32]

2. Other Pre Specified Outcome: Test Offer Rate
Description: The offer rate of the HIV test was defined as the proportion of enrolled study participants who were actually offered a test.
Time Frame: Assess on day subject enrolled into the study
Measure: Number; unit: participants
Arm/Group | Counselor | Provider
Number analyzed (Participants) | 2446 | 2409
participants | 1959 | 861
Statistical Analysis 1: Comparison: Counselor vs Provider; HIV test offered; Test type: Superiority or Other; p < 0.001, Chi-squared; Rate Difference (%) = 44, 95% CI 2-sided [42 to 47]

3. Other Pre Specified Outcome: Test Acceptance Rate
Description: Acceptance of the HIV test was defined as the proportion of study participants who received the HIV test among those offered the test.
Time Frame: Assess on day subject enrolled into the study
Population: Number of participants analyzed equals the number of participants offered a rapid HIV test. Many participants left the ED before the opportunity was available to offer the test.
Measure: Number; unit: participants
Arm/Group | Counselor | Provider
Number analyzed (Participants) | 1959 | 861
participants | 1382 | 643
Statistical Analysis 1: Comparison: Counselor vs Provider; HIV test accepted among patients offered; Test type: Superiority or Other; p = 0.02, Chi-squared; Rate Difference (%) = -4, 95% CI 2-sided [-8 to -1]

4. Primary Outcome: Linkage to Care of Newly Diagnosed HIV Infected Participants
Description: We define linkage to care as attendance at a first HIV clinic appointment where the following 3 events occur: 1) introduction to an HIV care primary provider; 2) receipt of confirmatory Western Blot HIV test results; and 3) phlebotomy for CD4 cell count and HIV RNA level.
Time Frame: Assessed within 8 weeks after receipt of reactive rapid HIV test results
Population: DSMB recommended the trial be ended early for likely inability to obtain this primary outcome. Thus the outcomes reported in paper are the secondary and other pre-specified outcomes listed.
Measure: Number; unit: participants
Arm/Group | Counselor | Provider
Number analyzed (Participants) | 2446 | 2409
participants
  Positive HIV Test | 0 | 7
  Linked to Care | 0 | 4

ADVERSE EVENTS:
Time Frame: 1 week after rapid HIV testing.
Arm/Group | Counselor | Provider
Serious Adverse Events (participants affected / at risk) | 0/1382 | 0/643
Other Adverse Events (participants affected / at risk) | 33/1382 | 14/643
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Counselor (N=1382) | Provider (N=643)
False-positive rapid test result (Investigations) | 27 (27) | 9 (9)
Subject did not follow-up after reactive test (Investigations) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes